CLINICAL TRIAL: NCT04167722
Title: The EXOPRO Study: How Does Prostate Cancer Metastasize? Understanding the Role of Exosomal Communication in Lean vs Obese Patients
Brief Title: How Does Prostate Cancer Metastasize? Studying the Role of Secreted Packages (Exosomes) From Fat Tissue in Lean and Obese Patients
Acronym: EXOPRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Experimental Cancer Medicine Centres (Other)
Responsible Party: Sponsor
Other Study IDs: 19HH5065
Record Dates: First submitted 2019-11-11; First posted 2019-11-19 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer; Obesity
Keywords: Prostate Cancer; Obesity; Exosomes
MeSH Terms: conditions — Prostatic Neoplasms; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Prostate cancer tissue, benign prostate tissue, peri-prostatic adipose tissue, omental adipose tissue, blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese patients: BMI > 25
  Interventions: Procedure: Robotic Radical Prostatectomy
- Lean patients: BMI < or = 25
  Interventions: Procedure: Robotic Radical Prostatectomy

INTERVENTIONS:
Procedure: Robotic Radical Prostatectomy — Routine NHS Radical Prostatectomy

SUMMARY:
The investigators will be collecting prostate and fat tissue from participants undergoing radical prostatectomy to culture and study in the laboratory.

DETAILED DESCRIPTION:
Both obesity and prostate cancer are major health problems in the UK, affecting 1 in 3 and 1 in 8 men respectively. Moreover, obesity increases the risk of developing aggressive disease and the risk of prostate cancer spreading. How this happens is not known. The investigators want to understand how fat cells communicate with prostate cancer cells. Investigators will be collecting prostate and fat tissue from radical prostatectomy participants for culture, in particular to look at exosome communication.

ELIGIBILITY:
Inclusion Criteria:

* All men undergoing radical prostatectomy at Charing Cross Hospital

Exclusion Criteria:

* Patients unable to consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Biological male only (can include transgender women)
Study Population: Obese vs lean patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Determine functional differences of peri-prostatic adipose tissue from lean vs obese patients on prostate cancer cell lines | Through to study completion, on average 3 years
  Proliferation, migration, invasion, apoptosis and epthelial-mesenchymal transition assays will be performed using isolated exosomes on prostate cancer cell lines
Identification of exosomal small RNAs transferred between human adipose tissue to prostate cancer cells lines | Through to study completion, on average 3 years
  Exosomal RNA transferred from human adipose tissue to prostate cancer cell lines will be isolated using a tagged magnetic bead isolation method and sequenced to identify transferred small RNAs
Assess how exosomal small RNAs from lean vs obese patients affect cancer regulation | Through to study completion, on average 3 years
  Prostate cancer cell lines will be treated with isolated exosomes, then parental and treated cells sequenced to identify differentially expressed RNA and underlying changes
Attempt to replicate functional changes observed | Through to study completion, on average 3 years
  Treatment of prostate cancer cell lines with microRNA mimics or inhibitors and comparison of changes with exosome treated cell lines

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Bevan, PhD, Principal Investigator — Imperial College London; Mathias Winkler, FRCS, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Charing Cross Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcomes will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 to 12 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Regulators will be required to sign a data access agreement.
URL: https://www.imperial.ac.uk/department-surgery-cancer/research/cancer/research-areas/clinical-trials/exopro-study/